CLINICAL TRIAL: NCT07383051
Title: Predictors of Successful Extubation of Pediatric Patients From Mechanical Ventilation With or Without Post Extubation High Velocity Nasal Insufflation
Brief Title: Randomized Clinical Trial for Predictors of Successful Extubation of Pediatric Patients From Mechanical Ventilation Either on High Velocity Nasal Insufflation or Simple Nasal Oxygen and Comparing the Outcome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Tarek Fayez Ali, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MD-299-2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Comparing the Outcome Between High Velocity Nasal Insufflation and Simple Oxygen After Successful Weaning From Mechanical Ventilation

STUDY DESIGN:
Intervention Model Description: comparing the outcome between High Velocity Nasal Insufflation and simple oxygen after successful weaning from mechanical ventilation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exubation of pediatric patients on High Velocity Nasal Insufflation (Experimental)
  Interventions: Device: Comparing the outcome of pediatric patients after successful weaning on either High Velocity Nasal Insufflation or simple oxygen; Device: comparing High Velocity Nasal Insufflation to simple oxygen after successful weaning of pediatric patients
- Exubation of pediatric patients on simple oxygen (Active Comparator)
  Interventions: Device: Comparing the outcome of pediatric patients after successful weaning on either High Velocity Nasal Insufflation or simple oxygen; Device: comparing High Velocity Nasal Insufflation to simple oxygen after successful weaning of pediatric patients

INTERVENTIONS:
Device: Comparing the outcome of pediatric patients after successful weaning on either High Velocity Nasal Insufflation or simple oxygen — A randomized clinical study is comparing between extubation on High Velocity Nasal Insufflation or simple nasal Oxygen ensuring that all patients had successful weaning predictors before extubation and comparing the outcome whether patient needed upgrading of oxygen support or reintubation within 48 hours, presence of respiratory distress or stridor post extubation, knowing mechanical ventilaton free days after extubation, time of complete weaning of oxygen support to room air and also morbidity and mortality.
Device: comparing High Velocity Nasal Insufflation to simple oxygen after successful weaning of pediatric patients — A randomized clinical study is comparing between extubation on High Velocity Nasal Insufflation or simple nasal Oxygen ensuring that all patients had successful weaning predictors before extubation and comparing the outcome whether patient needed upgrading of oxygen support or reintubation within 48 hours, presence of respiratory distress or stridor post extubation, knowing mechanical ventilaton free days after extubation, time of complete weaning of oxygen support to room air and also morbidity and mortality.

SUMMARY:
A randomized clinical trial about predictors of successful extubation of pediatric patients from mechanical ventilation either on High Velocity Nasal Insufflation or simple nasal oxygen and comparing the outcome

DETAILED DESCRIPTION:
A randomized clinical study is comparing between extubation on High Velocity Nasal Insufflation or simple nasal Oxygen ensuring that all patients had successful weaning predictors before extubation and comparing the outcome whether patient needed upgrading of oxygen support or reintubation within 48 hours, presence of respiratory distress or stridor post extubation, knowing mechanical ventilaton free days after extubation, time of complete weaning of oxygen support to room air and also morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 months and 13 years old with minimum weight 4kg
* Both sexes
* Patients on mechanical ventilation for at least 24 hours for any indication

Exclusion Criteria:

* Patients not ready for weaning from mechanical ventilation
* Contraindications to use of High velocity nasal insufflation
* Prolonged mechanical ventilation for more than 21 days

Ages: 2 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
comparing the need for reintubation within 48 hours afterr extubation using High Velocity Nasal Insufflation versus simple oxygen | 48 hours
  Successful extubation with no need for reintubation within 48 hours among pediatric ICU patients in those using High Velocity Nasal Insufflation versus simple oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Cairo University Cairo University, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt